CLINICAL TRIAL: NCT06829173
Title: A Phase 0/I Study to Assess the Safety and Tolerability of XRD-0394 in Combination With Radiation Therapy in Patients With High Grade Gliomas
Brief Title: Concurrent XRD-0394 With Radiation Therapy for High Grade Gliomas
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-01715
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: High-Grade Glioma
MeSH Terms: conditions — Glioma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pre-Surgery Dose-Escalation (Experimental): Patients with newly-diagnosed high grade gliomas (HGG) receiving neoadjuvant radiation therapy (RT) prior to surgical resection will be enrolled in the Pre-Surgical Dose-Escalation arm, at one of two dose levels:
  Participants enrolled at Pre-Surgical Dose Level 1 (DL1) will receive 160mg daily XRD-0394 on the days of radiation therapy before surgery.
  Participants enrolled at Pre-Surgery Dose Level 2 (DL2) will receive 300mg daily XRD-0394 on the days of radiation therapy before surgery.
  All patients enrolled in the pre-surgical dose escalation portion of the study will receive DL1 in the post-surgical dose-escalation portion of the study, but will not be enrolled in the Post-Surgery Dose Escalation arms for purpose of analysis.
  Interventions: Drug: XRD-0394; Radiation: Radiation Therapy; Procedure: Surgical Resection
- Cohort A: Post-Surgery Dose Escalation (Experimental): MGMT-methylated patients will be enrolled in Cohort A following surgical resection.
  Participants enrolled at Post-Surgery Dose-Level 1 (DL1) will receive 160 mg XRD-0394 administered twice weekly, concurrently with radiation therapy.
  Participants enrolled at Post-Surgery Dose-Level 2 (DL2) will receive 160 mg XRD-0394 administered three times weekly, concurrently with radiation therapy.
  Participants enrolled at Post-Surgery Dose-Level 3 (DL3) will receive 300 mg XRD-0394 administered three times weekly, concurrently with radiation therapy.
  Interventions: Drug: XRD-0394; Radiation: Radiation Therapy; Procedure: Surgical Resection
- Cohort B: Post-Surgery Dose Escalation (Experimental): MGMT-unmethylated patients will be enrolled in Cohort B following surgical resection.
  Participants enrolled at Post-Surgery Dose-Level 1 (DL1) will receive 160 mg XRD-0394 administered twice weekly, concurrently with radiation therapy.
  Participants enrolled at Post-Surgery Dose-Level 2 (DL2) will receive 160 mg XRD-0394 administered three times weekly, concurrently with radiation therapy.
  Participants enrolled at Post-Surgery Dose-Level 2 (DL3) will receive 300 mg XRD-0394 administered three times weekly, concurrently with radiation therapy.
  Interventions: Drug: XRD-0394; Radiation: Radiation Therapy; Procedure: Surgical Resection
- Cohort C: Dose-Escalation (No Surgery) (Experimental): Patients with recurrent high-grade glioma (HGG) will be enrolled in Cohort C.
  Participants enrolled at Dose-Level 1 (DL1) will receive 160 mg XRD-0394 administered twice weekly, concurrently with radiation therapy.
  Participants enrolled at Dose-Level 2 (DL2) will receive 160 mg XRD-0394 administered three times weekly, concurrently with radiation therapy.
  Participants enrolled at Dose-Level 2 (DL3) will receive 300 mg XRD-0394 administered three times weekly, concurrently with radiation therapy.
  Interventions: Drug: XRD-0394; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: XRD-0394 — Administered orally; small molecule dual inhibitor of ataxia telangiectasia mutated kinase (ATM) and DNA-PK.
Radiation: Radiation Therapy — For Cohort A and Cohort B, the neoadjuvant "boost" radiation dose is 1400cGy delivered over 7 fractions, and the adjuvant radiation dose is 5000cGy delivered over 25 fractions for a total dose of 6400cGy over 32 fractions, accounting for the treatment break between boost and adjuvant RT.
  For Cohort C, the radiation dose is 3500cGy delivered over 10 fractions.
Procedure: Surgical Resection — Resection of tumor tissue.
  Arms: Cohort A: Post-Surgery Dose Escalation; Cohort B: Post-Surgery Dose Escalation; Pre-Surgery Dose-Escalation

SUMMARY:
This is an open-label, dose-finding study of XRD-0394 in subjects with newly diagnosed and recurrent high grade gliomas receiving radiation therapy, with and without concurrent temozolomide based on O6-Methylguanine-DNA methyltransferase (MGMT) status for patients with newly diagnosed high grade gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* ≥18 years of age.
* For Cohorts A and B, radiographic diagnosis of high-grade glioma that is then confirmed with biopsy. Patients with established histologic diagnosis of high-grade glioma is able to enroll on the study without repeating biopsy.
* For Cohort C, histologic diagnosis of high-grade glioma is required to enroll on the study.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Subjects must have adequate liver and kidney function, defined as: Liver transaminase levels ≤2.5 × the upper limit of normal (ULN); total bilirubin ≤1.5 × ULN, except in subjects with Gilbert's Disease in whom total bilirubin ≤5 × ULN is allowed; OR Creatinine clearance ≥60 mL/min measured from a 24-hour urine collection or calculated based on the Cockcroft-Gault formula.
* Female subjects of childbearing potential and male subjects with female partners of childbearing potential must be willing to avoid pregnancy. Female subjects of childbearing potential who are undergoing RT or who are partners to male subjects in the study should avoid sexual activity or use a highly effective method of birth control during sexual intercourse. Acceptable, highly effective methods of birth control include intrauterine device (IUD)/intrauterine hormone releasing system (IUS), bilateral tube occlusion, vasectomized partner, combined (estrogen and progesterone containing) or progesterone-only hormonal contraceptives (oral, intravaginal, transdermal, injectable).
* Subjects receiving anti-glioma therapy are eligible if treatment can be held 14 days before the first XRD-0394 dose and resume a minimum of 5 days after completion of XRD-0394 (Cohort C only).
* Patient with recurrent tumor amendable to reirradiation and is at least 3 months from end of prior brain radiation therapy (Cohort C only)
* Subjects taking glucocorticoids before and during protocol treatment period will be included per the discretion of the investigator. Intake should be minimized before and during treatment.

Exclusion Criteria:

* Prior radiotherapy to the same region or prior anti-glioma systemic therapy in patients with newly diagnosed HGG (Cohorts A and B, not applicable for Cohort C)
* Subjects with bone marrow impairment as evidenced by hemoglobin <8.0 g/dL, neutrophil count <1.5 × 109/L, or platelets <100 × 109/L.
* History of difficulty swallowing, malabsorption or other chronic gastrointestinal disease or condition that may hamper compliance and/or absorption of XRD-0394, use of percutaneous endoscopic gastrostomy (PEG) tubes.
* Significant cardiac conduction abnormalities, including a history of long corrected QT (QTc) interval syndrome (>450 msec per Fridericia's formula) and/or pacemaker, or impaired cardiovascular function such as New York Heart Association classification >2 at screening.
* Participation in another investigational study of an unapproved drug or device or treatment with another ATM, deoxyribonucleic acid (DNA)-dependent protein kinase (DNA-PK), or ataxia-telangiectasia and Rad3-related (ATR) inhibitor within 28 days of the first dose of XRD-0394.
* Subjects who are pregnant or breast-feeding.
* Subjects with a QTc interval >450 msec (calculated using Fridericia's QT correction formula) at screening.
* Contraindication to temozolomide (Cohort A only)
* Severe headache, rapidly progressive neurologic decline, objective neurologic manifestations of uncal herniation, depressed level of consciousness
* Subjects receiving treatment with any drug that is a strong inhibitor or inducer of CYP3A4 enzyme activity or an inhibitor of BCRP within a minimum of 5 half- lives or 14 days prior to screening or during study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experience Dose-Limiting Toxicities (DLTs) | End of DLT Monitoring Period (Pre-surgical dose-escalation: Day 8; Cohort C: Day 44; Cohorts A & B: Day 108)
  Assessed among patients who receive at least one dose of the study drug and are evaluated for dose-limiting toxicities (DLTs).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to Year 3 Post-Enrollment
  Assessed among Cohorts A, B, and C only. Defined as the time from the start of treatment until the first documented disease progression or death.
Overall Survival (OS) | Up to Year 3 Post-Enrollment
  Assessed among Cohorts A, B, and C only. Defined as the time from treatment initiation until death from any cause.
Maximum Concentration (Cmax) of XRD-0394 in Resected Tumor Tissue | Day 8 (Day of Surgery)
  Assessed among Pre-Surgical Dose-Escalation participants only.
Area Under the Curve (AUC) of XRD-0394 in Resected Tumor Tissue | Day 8 (Day of Surgery)
  Assessed among Pre-Surgical Dose-Escalation participants only.
Time to Maximum Concentration (Tmax) of XRD-0394 in Resected Tumor Tissue | Day 8 (Day of Surgery)
  Assessed among Pre-Surgical Dose-Escalation participants only.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Yang, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Jonathan.Yang@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Jonathan.Yang@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.